CLINICAL TRIAL: NCT03415425
Title: Optimizing the Influenza Clinical Decision Support Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: QI-CDS
Record Dates: First submitted 2017-12-26; First posted 2018-01-30 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Clinical Decision Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): The current version of the alert will fire for this arm of the study.
  Interventions: Other: Current Version of the Influenza Alert
- Alert Iteration (Active Comparator): A modified version of the alert will fire for this arm of the study.
  Interventions: Other: Alternate Modifications of the Influenza Alert

INTERVENTIONS:
Other: Current Version of the Influenza Alert — Intervention includes the current version of the Influenza Alert that fires in the electronic medical record if the patient has not received the flu vaccination, as part of usual care.
  Arms: Usual Care
Other: Alternate Modifications of the Influenza Alert — Intervention includes various iterations of the Influenza Alert that fires in the electronic medical record if the patient has not received the flu vaccination.
  Arms: Alert Iteration

SUMMARY:
The proposed study aims to examine several iterations of the Influenza Best Practice Alert at NYU Langone Health. The goal is to increase ordering of the influenza vaccine through the alert.

ELIGIBILITY:
Inclusion Criteria:

* All NYU Langone Health inpatients eligible for the Influenza clinical decision support tool

Exclusion Criteria:

* N/A

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25881 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2023-10-07 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Alert Cancelation Rate | 2 months.
  Number of times alert fires in medical record within 2 Month period

SECONDARY OUTCOMES:
Vaccination Rate at Discharge | 2 months
  Number of vaccinations recorded in EMR within 2 Month period

CONTACTS AND LOCATIONS:
Overall Officials: Leora Horwitz, MD, MHS, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Austrian J, Mendoza F, Szerencsy A, Fenelon L, Horwitz LI, Jones S, Kuznetsova M, Mann DM. Applying A/B Testing to Clinical Decision Support: Rapid Randomized Controlled Trials. J Med Internet Res. 2021 Apr 9;23(4):e16651. doi: 10.2196/16651. PMID 33835035